CLINICAL TRIAL: NCT05091775
Title: The Evaluation of the Efficacy of Asacol (Mesalazine) Suppository on the Treatment of Diarrhea-Induced Acute Fissure in Post-Chemotherapy Cancer Patients - A Randomized Controlled Trial
Brief Title: The Efficacy of Asacol (Mesalazine) Suppository on the Treatment of Diarrhea-Induced Acute Fissure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Ghahramani, Clinical Associated professor of colorectal surgery, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 98-01-01-21181
Record Dates: First submitted 2021-04-27; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Fissure in Ano; Diarrhea
Keywords: Acute fissure; Diarrhea; Asacol
MeSH Terms: conditions — Fissure in Ano; Diarrhea

STUDY DESIGN:
Intervention Model Description: two groups seventy patients aged 18 to 65 years with diarrhea and subsequent acute fissure (with symptoms less than 6 weeks)
Who Masked: Care Provider
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard management of acute fissure(Diltiazem Jelly,supportive care,placebo suppository, sitz bath) (Placebo Comparator): Patients in the first group underwent for 14 consecutive days treatment with diltiazem gel 2 times a day, a basin of warm water 2 times a day and drink daily 8-12 a glass of water will be placed with a placebo suppository.
  Interventions: Drug: Asacol is used to treat and prevent mild to moderate acute fissure disease
- Intervention group (Asacol suppository, supportive care, placebo suppository, sitz bath) (Experimental): Patients in the second group or treatment group will be treated with diltiazem gel topically 3 times a day for 14 consecutive days, pelvis of warm water 2 times a day and drink daily 8-12 glasses of water plus Asacol anal suppository (mesalazine) are taken 1 piece every night.
  Interventions: Drug: Asacol is used to treat and prevent mild to moderate acute fissure disease

INTERVENTIONS:
Drug: Asacol is used to treat and prevent mild to moderate acute fissure disease — Comparison of two groups after 2 weeks in fissure wound healing, pain relief, pruritus, burning, bleeding, incontinence. Preliminary results of the study show the rate of fissure improvement 6 weeks after treatment, which is observed by clinical examination. Restoration is defined by complete epithelialization of the fissure site without scarring or residual cracks, and the secondary results will be a reduction in the amount of pain and other symptoms.
  Other Names: Mesalazine is used to treat and prevent mild to moderate acute fissure disease

SUMMARY:
Anal fissure define as a superficial tearing in mucosa on the anoderm surface distal to dentate line . The most important factor is hard stool passing with trauma to anal mucosa. But, diarrhea diarrhea has been another important etiology that happen after some conditions like gastroenteritis, laxative over use, during chemotherapy, and ulcerative colitis exacerbation . In these conditions, it seems the change of stool PH maybe the main reason of inflammation and ulcer in acute phase.

The treatment of acute is medical management with change in bowel habits and conservative therapy such as local lubricant, local vasodilator, and warm sitz bath to improve blood supply and wound healing.

This research clinical trial is designed to show the effect of Asacol suppository in the management of acute fissure due to diarrhea. The hypothesis of this research clinical trial has been referred to the cause of acute fissure ulcer because of diarrhea.

DETAILED DESCRIPTION:
The cases with acute anal fissure after diarrhea will included in this research clinical trial. They will be divided in two groups as an interventional group and control by blind randomization allocation. The interventional group will have received Asacol suppository 1 supp every night and Diltiazem jelly (standard management) twice per day. The control group will have received Diltiazem jelly and placebo suppository like interventional group. Both group will have used warm sitz bath with enough hydration for 10 days. Then the patients will have visited by another surgeon after 4 weeks to evaluate the healing of acute anal fissure. Pain will have performed if the patients can tolerate.

ELIGIBILITY:
Inclusion Criteria:

For age between 18 and 65 years are the presence of acute anal fissure (with symptoms less than 6 weeks) following chronic diarrhea and subsequent fissure.

Exclusion Criteria:

* Recurrent fissure with skin appendage.
* Long history of constipation.
* Use of immunosuppressive drugs or corticosteroids.
* Inflammatory bowel disease such as Crohn's disease and ulcerative colitis.
* Pregnancy.
* Grade 3 and 4 hemorrhoids.
* Neurological disease.
* Obsessive-compulsive disorder.
* Previous history of anal surgery
* Skin diseases such as eczema and psoriasis.
* Sexually transmitted infections, tuberculosis.
* Mucosal prolapse.
* Anal fistula and pelvic radiotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Acute anal fissure after diarrhea. Standard management of acute fissure (Diltiazem Jelly, supportive care, placebo suppository, sitz bath) | 2 weeks
  bleeding anal fissure. After 2weeks the patients will visit. The score of pain, burning sensation, bleeding and improvement will be recorded in two groups.
  Score of pain with visual analog scale (VAS) is a tool widely used to measure pain; Scale (0-10) that higher grade means higher pain. Burning sensation (yes, no) and bleeding (yes, no) and improvement (yes, no) will be recorded

SECONDARY OUTCOMES:
Acute anal fissure after diarrhea. Intervention group (Asacol suppository, supportive care, placebo suppository, sitz bath) | 3 months
  need surgery or botox injection. Both group including 70 patients that will visit after 2 weeks for evaluating heading acute fissure by history and physical examination.
  Bleeding(decrease/increase) Pruritus(decrease/increase) Wound healing (according to surgeon evaluation)

CONTACTS AND LOCATIONS:
Locations (1):
- Leila Ghahramani, Shiraz, Fars, Iran